CLINICAL TRIAL: NCT04242303
Title: Evaluation of the Effectiveness of a Technique Based on Inertial Sensors vs the Conventional Technique for the Execution of the Bone Resections in Primary Total Knee Arthroplasty: a Controlled Randomized Trial
Brief Title: Effectiveness of Inertial Sensors vs the Conventional Technique for the Execution of the Bone Resections in Primary TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TKA_EM2
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: The patients will be divided into 2 groups, based on the alignment technique used Total number of patients involved: 180 (90 Group A Patients: EM Technique), (90 Group B Patients: IM Technique) Total number of centers involved: 3 Patients per Center: 30 Group A Patients, 30 Group B Patients
Who Masked: Outcomes Assessor
Masking Description: The evaluation of the results obtained will be carried out blindly by an examiner with adequate clinical skills to carry out the evaluation and who does not take part in the operational phases of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EM Technique (Experimental): use of extramedullary technique by means of inertial sensors for the execution of femoral cuts
  Interventions: Procedure: Total knee replacement
- IM Technique (Active Comparator): Use of conventional intramedullary technique for the execution of femoral cuts
  Interventions: Procedure: Total knee replacement

INTERVENTIONS:
Procedure: Total knee replacement — Total knee arthroplasty using standard anterior approach. In the EM group, inertial sensor will be used to perform femoral bone cuts.
  In the IM group, conventional intramedullary nail will be used as reference to perform femoral bone cuts.

SUMMARY:
Comparison of surgical technique for the execution of bone resections in total knee arthroplasty.

Used technique are: a non-invasive extramedullary technique (EM technique) based on the use of inertial sensors for cutting guides positioning and conventional technique (IM technique), based on the use on intramedullary stem.

Our hypothesis is that the EM technique based on the use of inertial sensors leads to a reduction in the number of outliers equal to or greater than 20% compared to the outliers obtained with the conventional technique.

DETAILED DESCRIPTION:
Comparison of surgical technique for the execution of bone resections in total knee arthroplasty.

Used technique are: a non-invasive extramedullary technique (EM technique) based on the use of inertial sensors for cutting guides positioning and conventional technique (IM technique), based on the use on intramedullary stem. A study was carried out at the Rizzoli Orthopedic Institute in 2016 to compare non-invasive extramedullary technique (EM technique) and conventional technique (IM technique). Starting from the results obtained in the previous study, the objective of this study is to deepen the investigations to evaluate the effectiveness of the EM technique compared to the conventional IM technique.

The patients involved in the study will be divided into two groups based on the alignment technique used (EM technique and IM technique).

The results obtained will be measured on postoperative panoramic radiographs at discharge, assessing the overall alignment of the limb and the individual femoral and tibial components in terms of accuracy and repeatability according to a defined measurement protocol.

Primary endpoint:

- reduction in the number of cases in which the alignment error on the coronal plane is greater than 3°of error (outlier). Our hypothesis is that the EM technique based on the use of inertial sensors leads to a reduction in the number of outliers equal to or greater than 20% compared to the outliers obtained with the conventional technique.

Secondary endpoints:

* the reduction of the variation in hemoglobin levels during hospitalization. Our hypothesis is that the EM technique leads to a reduction in the maximum variation of hemoglobin levels during the hospitalization period compared to the IM technique equal to or greater than 1g / dl
* reduction of alignment errors of the femoral and tibial resections obtained with the EM technique and with the IM technique on the sagittal plane. In particular, the experimental hypothesis is that in the EM technique group, values of alignment of the implant with respect to the femoral and tibial mechanical axis on the sagittal plane are not significantly lower than those obtained with the standard technique but with a reduction in the standard deviation in the EM group compared to the IM group.
* reduction of the period of hospital stay in the EM group compared to the group operated with the standard technique.
* inter-operator variability in the EM group Randomized controlled multicenter prospective study. The evaluation of the results obtained will be blinded by an examiner with adequate clinical skills and who does not take part in the operational phases of the study.

Duration: 36 months The patients will be divided into 2 groups, based on the alignment technique used Total number of patients involved: 180 (90 Group A Patients: EM Technique), (90 Group B Patients: IM Technique) Total number of centers involved: 3 Patients per Center: 30 Group A Patients, 30 Group B Patients Patients will be randomized. The randomization list will be generated using the website www.randomization.com. This list will be kept at the Operative Unit Orthopedic and Traumatological Clinic 2nd and will not be visible to the investigators involved The evaluation of the results obtained will be carried out blindly by an examiner with adequate clinical skills to carry out the evaluation and who does not take part in the operational phases of the study.

For both groups of patients, the results obtained will be measured on postoperative panoramic radiographs performed at discharge, assessing in terms of accuracy and repeatability.

Finally, within Group A, the inter-operator variability of the measurement of the final femoral and tibial alignment obtained using the Blant & Altman analysis method will be assessed

The study involves the collection of data in three different phases:

Preoperative phase:

* Panoramic radiography under weight-bearing of the lower limbs in A-P and radiography of the knee in lateral projection
* laboratory value of hemoglobin

Intraoperative phase:

* Time of application of the ischemic snare;
* Surgery time;
* Final femoral and tibial alignment. In Group A the acquisition is repeated 2 times by two operators.
* Number of repetitions of distal femoral and tibial resections;
* Possible administration of blood products;
* Blood loss;

Post-operative phase

* Panoramic X-ray under weight-bearing of the lower limbs in A-P and knee radiography in lateral projection (at discharge)
* laboratory value of the patient's hemoglobin on each day until the date of discharge
* possible administration of blood products
* hospitalization times All data will be collected in a data collection form associated with the patient.

The preoperative and postoperative radiographs (made anonymous) and the data collection form will be sent to the coordinating center which will carry out the measurements.

From the literature it emerges that in order to detect a difference between the two techniques of 20% on the number of outliers (alignment of the components >±3°on the coronal plane) with an alpha type error (level of significance) equal to 0.05 and a power of at least 0.8, the minimum number of samples needed per group is 82 cases. Considering a 10% drop out, a sample of 90 cases per group is expected (divided into 3 centers for a total of 30 cases per group in each center)

ELIGIBILITY:
Inclusion Criteria:

* patients candidated for total knee arthroplasty
* hip mobility range of at least 30 °
* BMI <35kg / m2
* Aged between 40 and 80 years

Exclusion Criteria:

* ipsilateral hip arthrodesis or ankylosis
* non-perforable femoral medullary canal
* 165 °<HKA <195 °
* BMI> 35kg / m2

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Reduction in the number of cases in which the alignment error on the coronal plane is greater than 3°of error (outlier). | 22 months
  * HKA alignment on the coronal plane (medial angle between the femoral mechanical axis and the tibial mechanical axis)
  * coronal femoral angle (medial angle between the femoral mechanical axis and the tangent to the distal condyles of the femoral prosthetic component
  * tibial coronal angle (medial angle between the tibial mechanical axis and the tangent to the proximal profile of the tibial component) The number of patients with an HKA angle such that 180°-3°> HKA> 180°+ 3°or 180°-2°> HKA> 180°+ 2°will also be evaluated

SECONDARY OUTCOMES:
Reduction of the variation in hemoglobin levels during hospitalization. | 22 months
  The maximum variation of hemoglobin during the period of hospitalization will also be assessed within each group by comparing the hemoglobin value at the time of hospitalization with the hemoglobin values during the post-operative hospital stay
Reduction of alignment errors of the femoral and tibial resections obtained with the EM technique and with the IM technique on the sagittal plane | 22 months
  Sagittal femoral angle (angle between the mechanical femoral axis on the sagittal plane and the distal femoral resection plane) Tibial slope (angle between the tibial mechanical axis on the sagittal plane and the tangent to the proximal profile of the tibial component)
Reduction of the period of hospital stay in the EM group compared to the group operated with the standard technique | 22 months
  Hospital stay will be measured in day of hospitalization
Inter-operator variability in the EM group | 22 months
  The inter-operator variability of the measurement of the final femoral and tibial alignment obtained using the Blant & Altman analysis method will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Maria Marcheggiani Muccioli, MD, PhD, Principal Investigator — IRCCS Rizzoli Orthopedic Institute
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No